CLINICAL TRIAL: NCT05747404
Title: The FUnctional TricUspid REgurgitation by 3D EChocardiography Cooperative Study
Acronym: FUTURE 3D
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C040
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Heart Valve Incompetence; Echocardiography, Transthoracic
Keywords: Functional tricuspid regurgitation; Three-dimensional echocardiography; Doppler echocardiography; Right ventricular function; Right atrial function
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Functional tricuspid regurgitation: Patients with functional tricuspid regurgitation
  Interventions: Diagnostic Test: Echocardiography
- Control subjects: Healthy volunteers

INTERVENTIONS:
Diagnostic Test: Echocardiography — - Develop new parameters of FTR severity that take into account the lower momentum of the tricuspid regurgitant jet (compared with the mitral regurgitation jet), the complex anatomy of the regurgitant orifice, and both the intra-beat and respiratory variation of the regurgitant volume
  Groups: Functional tricuspid regurgitation

SUMMARY:
Prospective, multicenter, observational study to enroll consecutive patients with functional tricuspid regurgitation (FTR) with the primary aim to:

* Use patients' outcomes as a reference to try to define the threshold values for the different grades of FTR severity; and secondary aims to:
* Use 3D echocardiography to assess the relationships among the geometry (size and shape) of the right ventricle, right atrium, tricuspid annulus, and tricuspid leaflets according to the underlying cardiac condition (i.e., atrial fibrillation, pulmonary hypertension, right ventricular cardiomyopathy, congenital heart diseases, etc.)
* Assess the accuracy, and incremental diagnostic and prognostic value of a new software package to measure tricuspid annulus and valve geometry
* Develop new parameters of FTR severity that take into account the lower momentum of the tricuspid regurgitant jet (compared with the mitral regurgitation jet), the complex anatomy of the regurgitant orifice, and both the intra-beat and respiratory variation of the regurgitant volume
* Test the hypothesis that there is no actual grading but a continuum of increased risk of adverse outcome with the increase of FTR severity, and we need robust quantitative metrics (for example, the regurgitant fraction - currently not included in guidelines - which takes into account the right ventricular volume and function) more than grading schemes to assess the severity of the diseases and the effect of treatments
* Test the hypothesis that the relationship between FTR severity and the outcome may be different according to the underlying cardiac condition (i.e., atrial fibrillation, pulmonary hypertension, right ventricular cardiomyopathy, congenital heart diseases, post-cardiac surgery, etc.) as this will affect the timing for interventions

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years,
* signed informed consent to be part of this study,
* no pregnancy,
* the presence of at least one of the following cardiac conditions: a. Permanent atrial fibrillation b. Pulmonary arterial hypertension c. Left heart diseases with increased postcapillary pressure d. Right ventricular cardiomyopathy e. Right ventricular infarction f. Chronic thromboembolic pulmonary embolism g. Congenital diseases with right ventricular volume overload (atrial septal defect, interventricular septal defect, pulmonary regurgitation) h. Previous left heart valve surgery I. Good enough acoustic window and patient cooperation to obtain 3D echo data sets of the right ventricle, right atrium and tricuspid valve with a minimum temporal resolution of 20 vps l. Availability for clinical and echocardiography follow-up

Exclusion Criteria:

* Unwillingness to be part of the study
* Primary tricuspid valve disease
* Patient already scheduled for tricuspid valve repair/replacement
* Cardiac pacemaker, ICD or CRT leads
* Poor acoustic window
* Impossibility of left lateral decubitus position
* Extreme heart rates (<50 or >100 bpm)
* Previous LVAD implantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with at least mild functional tricuspid regurgitation and good apical acoustic window
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2027-04-21 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint | 5 years
  death from any cause and hospitalization for heart failure

OTHER OUTCOMES:
Right heart remodeling in various cardiac conditions affecting the right heart | 5 years
  Use 3D echocardiography to assess the relationships among the geometry (size and shape) of the right ventricle, right atrium, tricuspid annulus and tricuspid leaflets according to the underlying cardiac condition (i.e. atrial fibrillation, pulmonary hypertension, right ventricular cardiomyopathy, congenital heart diseases etc.)
3D echo software validation | 1 year
  Assess the accuracy, and incremental diagnostic and prognostic value of a new software package to measure tricuspid annulus and valve geometry
Improve grading of FTR | 2 years
  Develop new parameters of FTR severity that take into account the lower momentum of the tricuspid regurgitant jet (compared with the mitral regurgitation jet), the complex anatomy of the regurgitant orifice, and bot the intra-beat and respiratory variation of the regurgitant volume
Clinical significance of categorical grading | 5 years
  Test the hypothesis that there is no actual grading, but a continuum of increased risk of adverse outcome with the increase of FTR severity and we need robust quantitative metrics (for example the regurgitant fraction - currently not included in guidelines - which takes into account the right ventricular volume and function) more than grading schemes to assess the severity of the diseases and the effect of treatments
Define different phenotypes of FTR | 5 years
  Test the hypothesis that the relationship between FTR severity and outcome may be different according to the underlying cardiac condition (i.e. atrial fibrillation, pulmonary hypertension, right ventricular cardiomyopathy, congenital heart diseases, post-cardiac surgery etc.) as this will affect the timing for interventions

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Badano, MD, Ph.D., Study Director — Istituto Auxologico Italiano, IRCCS
Locations (4):
- Italy (2):
  - Istituto Auxologico Italiano, IRCCS, Milan
  - University of Padova, Padua
- Romania (2):
  - University of Medicine and Pharmacy Carol Davila, Bucharest
  - University of Medicine and Pharmacy of Craiova, Craiova

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request